CLINICAL TRIAL: NCT07179783
Title: Phase II Study of the Combination of Sacituzumab Tirumotecan(SKB264)and Tagitanlimab (KL-A167) in the Treatment of Aggressive Variant Prostate Cancer (AVPC) and Neuroendocrine Prostate Cancer (NEPC)
Brief Title: Sacituzumab Tirumotecan in Combination With Tagitanlimab in the Treatment of Aggressive Variant Prostate Cancer (AVPC) and Neuroendocrine Prostate Cancer (NEPC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Second Hospital (Other)
Collaborators: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-KL-A167-AVPC/NEPC-01
Record Dates: First submitted 2025-09-08; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer (Adenocarcinoma); Prostate Cancer Metastatic Castration-Resistant; Prostate Adenocarcinoma With Neuroendocrine Differentiation
Keywords: NEPC; AVPC; TROP2; PD-L1
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — 18-O-demethylcervinomycin A2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SKB264-KL-A167 Treatment Group (Experimental): This treatment group will receive a combination therapy of SKB264 and KL-A167.
  Interventions: Drug: Sacituzumab Tirumotecan; Drug: Tagitanlimab

INTERVENTIONS:
Drug: Sacituzumab Tirumotecan — Drug reduction will be implemented according to the research plan.
  Other Names: SKB264; Sac-TMT; MK-2870
Drug: Tagitanlimab — Treatment with Sacituzumab Tirumotecan (SKB264, 5mg/kg IV d1 Q2W) and Tagitanlimab (KL-A167 , 900mg IV d1 Q2W) until confirmed by the investigator as imaging disease progression, intolerable toxicity, subject's request to terminate treatment, or other treatment termination criteria specified in the protocol (based on the first patient), with a maximum treatment duration of 24 months for Tagitanlimab. Drug reduction will be implemented according to the research plan.
  Other Names: KL-A167

SUMMARY:
This study is a prospective, single arm II clinical trial. The main objective of the study is to evaluate the efficacy and safety of the combination of Sacituzumab Tirumotecan (SKB264) and Tagitanlimab (KL-A167) in the treatment of AVPC (aggressive variant prostate cancer) and NEPC (neuroendocrine prostate cancer).

DETAILED DESCRIPTION:
More than 60% of newly diagnosed cases of prostate cancer in China are in the middle and late stages, with an overall poor prognosis. Prostate cancer is AVPC (aggressive variant prostate cancer) and NEPC (neuroendocrine prostate cancer), two highly invasive and poorly prognosis non androgen receptor driven subtypes of prostate cancer. The overall prognosis of advanced AVPC and NEPC is poor, with a median OS of only 7-20 months after diagnosis. At present, there is a lack of a unified standard protocol for drug treatment of AVPC and NEPC. The recommended treatment plan in the diagnosis and treatment guidelines is mainly platinum based chemotherapy, as the behavior of AVPC and NEPC is similar to that of small cell lung cancer, and can be treated according to the guidelines for small cell lung cancer.More research is still underway on the use of immunotherapy combined with chemotherapy for advanced AVPC/NEPC. This study is a prospective, single arm II clinical trial. The main objective of the study is to evaluate the efficacy and safety of the combination of Sacituzumab Tirumotecan (SKB264) and Tagitanlimab (KL-A167) in the treatment of advanced AVPC and NEPC.The above research suggests that immunotherapy combined with chemotherapy has further exploration value in advanced AVPC/NEPC.

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of signing the informed consent form is ≥ 18 years old;
2. AVPC or NEPC diagnosed based on recent histological and/or clinical criteria;
3. Having received one or two second-generation anti androgen therapies in the past, previous use of docetaxel for castration resistant prostate cancer (CRPC) is allowed, and the use of other chemotherapy is not allowed;
4. The progression of prostate cancer in the subjects within 6 months prior to screening shall be determined by the researcher through one of the following methods:

   PSA is evaluated by local laboratories, and PSA progression is defined as at least two increases in PSA levels at intervals of ≥ 1 week, with a screening PSA value of ≥ 2 ng/ml.

   • Soft tissue imaging disease progression determined based on PCWG modified RECIST 1.1 or RECIST 1.1 criteria, regardless of PSA progression.

   The imaging disease progression of bones is defined as the appearance of two or more new bone lesions in bone scans, regardless of PSA progression.
5. Subjects who have not undergone past surgery must be using and voluntarily continue to use luteinizing hormone releasing hormone (LHRH) agonists throughout the entire study treatment period;
6. According to RECIST v1.1, there should be at least one measurable lesion, and previously irradiated lesions should not be selected as target lesions; Subjects with only skin or bone lesions are not eligible for inclusion;
7. Within 7 days prior to administration, the physical fitness status score of the Eastern Cooperative Oncology Group (ECOG) in the United States was 0 or 1;
8. Expected survival period ≥ 12 weeks;
9. Having sufficient organ and bone marrow function (without receiving blood transfusion, recombinant human thrombopoietin or colony-stimulating factor therapy within 2 weeks prior to administration), defined as follows:

   1. Blood routine: neutrophil count (NEUT #) ≥ 1.5 × 109/L; platelet count (PLT) ≥ 100 × 109/L; hemoglobin ≥ 90 g/L;
   2. Liver function: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN; For subjects with liver metastasis at baseline, ALT and AST should be ≤ 5 × ULN; Albumin ≥ 30g/L; Total bilirubin (TBIL) ≤ 1.5 × ULN;
   3. Renal function: creatinine clearance rate ≥ 50 ml/min (calculated using the standard Cockcroft Gault formula);
   4. Coagulation function: International normalized ratio (INR), activated partial thromboplastin time (APTT), and prothrombin time (PT) ≤ 1.5 × ULN;
10. For subjects whose partners have fertility potential, they must agree to take effective medical contraceptive measures within 6 months from the signing of the informed consent form until the last administration (see Annex 2 for details);
11. The subjects voluntarily joined this study, signed an informed consent form, and were able to comply with the visit and related procedures specified in the protocol.

Exclusion Criteria:

1. Previously received any of the following treatments (including in the context of adjuvant or neoadjuvant therapy):

   1. Targeted treatment of TROP2;
   2. Any drug therapy containing targeted topoisomerase I, including antibody conjugated drug (ADC) therapy;
   3. Immune checkpoint inhibitors (such as anti-PD-1/L1 antibodies, anti-CTLA-4 antibodies, etc.), immune checkpoint agonists (such as ICOS, CD40, CD137, GITR, OX40 antibodies, etc.), immune cell therapy, and any other treatment targeting the tumor immune mechanism;
2. Those who require the use of strong inhibitors or inducers of cytochrome P450 3A4 enzyme (CYP3A4) within 2 weeks prior to the first administration and during the study period (strong inhibitors or inducers of CYP3A4 are not allowed in this study, and representative drugs of CYP3A4 strong inhibitors or inducers are listed in Appendix 7); All subjects must avoid the concurrent use of any drugs, herbal supplements, and/or intake of such foods known to induce CYP3A4 as much as possible;
3. Subjects with central nervous system (CNS) metastases known to have meningeal metastases, brainstem metastases, spinal cord metastases and/or compression, active or untreated conditions. For subjects with brain metastases who have received local treatment in the past, if they have been clinically stable for at least 4 weeks before medication and have not required the use of glucocorticoids or anticonvulsants for at least 14 days, they are allowed to be enrolled;
4. Suffering from other malignant tumors within 3 years before administration (excluding tumors that have been cured through local treatment, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, cervical carcinoma in situ, etc.);
5. There are any of the following cardiovascular diseases or cardiovascular risk factors:

   1. Within 6 months prior to administration, if there is a myocardial infarction, unstable angina, acute or persistent myocardial ischemia, grade 3 or 4 heart failure (according to the New York Heart Association (NYHA) classification), symptomatic or poorly controlled severe arrhythmia, cerebrovascular accident, transient ischemic attack, or other serious cardiovascular and cerebrovascular diseases;
   2. Previous history of myocardial diseases such as myocarditis, primary cardiomyopathy, and specific cardiomyopathy;
   3. Any deep vein thrombosis (if stabilized for ≥ 2 weeks with low molecular weight heparin or similar efficacy drugs), peripheral arterial thromboembolic events, pulmonary embolism, or other serious thromboembolic events within 3 months prior to administration;
   4. Major vascular diseases that may endanger life or require surgery within 6 months prior to administration, such as aortic aneurysm, aortic dissection aneurysm, etc;
6. According to researchers' assessment, uncontrolled systemic diseases:

   1. Poor control of diabetes (fasting blood glucose ≥ 10 mmol/L for two consecutive times);
   2. Poor control of hypertension (systolic blood pressure>160 mmHg and/or diastolic blood pressure>100 mmHg);
   3. Presence of pleural effusion, pericardial effusion, or ascites with clinical symptoms or requiring repeated drainage (>once per week);
7. History of (non infectious) interstitial lung disease (ILD) or non infectious pneumonia requiring steroid treatment, current ILD or non infectious pneumonia, or suspected ILD or non infectious pneumonia that cannot be excluded by imaging examination during screening;
8. Clinical severe lung damage caused by concurrent lung diseases, including but not limited to any underlying lung disease (such as pulmonary embolism, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion, etc. within 3 months before administration) or any autoimmune, connective tissue, or inflammatory disease that may affect the lungs (i.e. rheumatoid arthritis, Sjogren's syndrome, sarcoidosis, etc.), or previous total pneumonectomy;
9. Subjects with active chronic inflammatory bowel disease, gastrointestinal obstruction, severe ulcers, gastrointestinal perforation, abdominal abscess, or acute gastrointestinal bleeding;
10. Individuals with bleeding tendencies such as acute gastrointestinal bleeding, persistent bleeding disorders, or coagulation dysfunction;
11. The toxicity of previous anti-tumor treatments has not yet recovered to ≤ level 1 (evaluated based on NCI CTCAE v5.0) or the levels specified in the inclusion and exclusion criteria (excluding toxicity judged by researchers to be of low safety risk such as hair loss and fatigue).
12. Suffering from active autoimmune diseases that require systemic treatment within the past two years (including but not limited to: autoimmune hepatitis, uveitis, enteritis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, etc.), systemic treatment includes drugs to improve the condition, immunosuppressants, systemic corticosteroid administration (>10 mg/day prednisone or equivalent drugs), etc. Hormone replacement therapy, such as thyroid hormone, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency, is not considered a systemic treatment; Subjects who received systemic corticosteroid treatment with>10 mg/day prednisone or other immunosuppressive drugs within 2 weeks prior to administration.
13. Known active pulmonary tuberculosis. Subjects suspected of having active pulmonary tuberculosis need to undergo clinical examination for exclusion;
14. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
15. Accompanied by ≥ grade 2 peripheral neuropathy;
16. Active hepatitis B [hepatitis B surface antigen (HBsAg) is positive, and HBV-DNA detection is required; HBV-DNA ≥ 500 IU/mL or higher than the lower limit of detection, whichever is higher] or hepatitis C (positive for hepatitis C antibodies and HCV-RNA above the lower limit of detection). Note: HBsAg positive subjects are required to receive anti hepatitis B virus treatment during the study treatment;
17. Human immunodeficiency virus (HIV) test is positive or there is a history of acquired immunodeficiency syndrome (AIDS); Known active syphilis infection;
18. Known allergies to the investigational drug or any of its components, and a history of severe hypersensitivity reactions to other biological agents;
19. Individuals who have undergone major surgery within 4 weeks prior to administration or are expected to undergo major surgery during the study period;
20. Serious infection occurred within 4 weeks prior to administration, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia; Within 2 weeks prior to administration, there is an active infection that requires systemic anti infective treatment;
21. A recorded history of severe dry eye syndrome, severe meibomian gland disease and/or meibomian inflammation, or corneal diseases that hinder delayed corneal healing;
22. Have received non-specific immunomodulation therapy (including but not limited to interferon and IL-2), traditional Chinese patent medicines and simple preparations preparations with approved anti-tumor indications, etc. within 2 weeks before administration;
23. Received a live vaccine within 30 days prior to administration, or planned to receive a live vaccine during the study period; During the screening process before administration, the condition rapidly deteriorates, such as significant changes in physical fitness status;

25) Suffering from local or systemic diseases caused by non malignant tumors, or diseases or symptoms secondary to tumors, which can lead to higher medical risks and/or uncertainty in survival evaluation, such as tumor like leukemia reactions, cachexia manifestations, etc; 26) Any condition that the researcher deems to interfere with the evaluation of the investigational drug, the safety of the subjects, or the interpretation of the research results, or any other condition that the researcher deems unsuitable for participation in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective Response Rate (ORR) assessed according to the evaluation criteria for the efficacy of solid tumors (RECIST v1.1)/ Prostate Cancer Clinical Trials Working Group(PCWG3).

SECONDARY OUTCOMES:
Progression Free Survival(PFS) | From treatment administration up to a maximum duration of 24 months.
  The time from the beginning of the patient's treatment to the disease progression or death for any reason. Based on RECIST criteria v1.1/ PCWG3.
Duration of Response(DOR) | Through study completion, an expected average of 24 months.
  Duration of Response, from the first time the evaluation results meet CR or PR criteria to the observation of PD or death.
Disease Control Rate (DCR) | From treatment administration up to a maximum duration of 24 months.
  The proportion of subjects with complete response (CR) and partial response (PR) and stable disease (SD) in total subjects after the last subject participating in.
Overall Survival(OS) | From treatment administration up to a maximum duration of 24 months.
  Time from start of treatment to death due to any cause.
Percentage of Participants With Adverse Events (AEs) | Up to approximately 24 months.
  Number of participants with adverse effects of treatment. Frequency and severity of adverse effects of treatment as assessed by NCI CTCAE v5.0.

OTHER OUTCOMES:
Exploring predictive effectiveness indicator | Up to approximately 24 months.
  Explore potential biomarkers for predicting therapeutic efficacy, including but not limited to immune related indicators such as PD-L1, TILs, lymphocyte subsets, and TROP2 expression.

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Wang, Ph.D, Study Chair — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
After the experiment is completed, the data maybe shared after academic publication.